CLINICAL TRIAL: NCT00591032
Title: Development of Rational and Standardized Diagnostics and Staging for a Differentiated Risk Stratification of Non-thyroidal Illness Syndrome
Brief Title: Approach to a Quantitative Follow-up of Non-thyroidal Illness Syndrome
Acronym: AQUA FONTIS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Wissenschaftskommission des Universitaetsklinikums Bergmannsheil (Unknown); Private Sponsor (Chantal C. Guilhemotonia-Urban) (Unknown)
Responsible Party: Principal Investigator, PD Dr. Johannes W. Dietrich, MD, Senior consultant endocrinologist, Ruhr University of Bochum
Other Study IDs: 2006-Innere-565; 2848 (Other: Ethics Committee ID); U1111-1122-3245 (Registry Identifier: WHO ICTRP Universal Trial Number (UTN)); DRKS00003152 (Registry Identifier: DRKS (German Clinical Trials Register))
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Euthyroid Sick Syndromes; Non-thyroidal Illness Syndrome; Low T3 Syndrome; TACITUS
Keywords: Critical illness; Euthyroid sick syndromes; Intensive care; Non-thyroidal illness syndrome; Low-T3 syndrome
MeSH Terms: conditions — Euthyroid Sick Syndromes; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Kryobase with serum and urine samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
AQUA FONTIS is a unicentric, multidisciplinary, prospective cross-section and longitudinal study that aims at the development of a more clear-cut diagnostic definition and classification of non-thyroidal illness syndrome (NTIS).

DETAILED DESCRIPTION:
Detailed Description:

Non-thyroidal illness syndrome (NTIS), also referred to as euthyroid sick syndrome (ESS) or thyroid allostasis in critical illness, tumors, uremia and starvation (TACITUS), is a complex endocrine condition that may occur in critically ill patients. It is associated with significantly increased morbidity and mortality.

NTIS is characterised by three components that may occur single or in combination:

1. central hypothyroidism (transient thyrotropic insufficiency)
2. impaired protein binding of thyroid hormones and
3. reduced formation of T3 and increased conversion to rT3 (low-T3-syndrome).

Despite of long lasting research to some of its details NTIS is still poorly characterized in an integrative view. Additionally, it lacks a clinically usable classification.

Given the fact that patients with NTIS are faced with poor prognosis, several studies have been conducted in the past evaluating the question of possible treatment. However, they didn't yield unambiguous results, maybe due to the fact that these studies did not differentiate among the distinct components of NTIS.

Therefore, this study is intended to develop a clear-cut definition and classification of NTIS in order to set a foundation for future therapeutic studies.

This study recruits critically ill patients treated in medical and surgical intensive care units of the Bergmannsheil University hospitals for evaluation of integrative thyrotropic control and follow-up. From these data the correlation of individual prognosis with laboratory-defined components of NTIS will be determined.

This project is intended to:

1. deliver a prognostical aid by providing a differentiated classification,
2. to contribute to a standardised, rational and inexpensive diagnostical procedure and
3. to lay the foundation for future therapeutic trials by identifying subgroups that may benefit from therapy.

ELIGIBILITY:
Inclusion Criteria:

* Severe illness requiring intensive care
* Stay of at least 24 hours at the ICU

Exclusion Criteria:

* Substituted hypothyroidism or substitution in case of thyroid carcinoma
* Hyperthyroidism that is treated with thyrostatic agents and exhibits a THS level not below the reference region
* Manifest AIDS disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients treated at three intensive care units of the Bergmannsheil university hospitals and that comply with the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2007-05; Primary Completion 2017-11-30 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the significance of an innovative physiological index approach (SPINA) in differential diagnosis between NTIS and latent thyrotoxicosis. | Three weeks after admission to ICU (evaluation point 1.5) and additionally on day of discharge from the hospital (evaluation point 1.999)
  Diagnostic accuracy (sensitivity, specificity and AUCs of ROC analysis) of the thyroid's calculated secretory capacity (GT) for differentiation between NTIS and subclinical hyperthyroidism.

SECONDARY OUTCOMES:
Correlation of variables that quantify distinct components of NTIS with independent predictors of evolution, survival or pathophysiological condition and influencing or disturbing factors like medication. | 24 hours (evaluation point 1.1), 72 hours (evaluation point 1.2) and further on weekly (evaluation points 1.3 to 1.5) after admission to the intensive care unit up to the day of discharge from hospital (evaluation point 1.999)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes W Dietrich, M.D., Principal Investigator — Medizinische Klinik I, Universitätsklinikum Bergmannsheil, Ruhr-Universität Bochum; Steffen Hering, M.D., Study Director — Diabetes-Zentrum, Mathias-Spital Rheine; H H Klein, M.D., Study Chair — Medizinische Klinik I, Universitätsklinikum Bergmannsheil, Ruhr-Universität Bochum
Locations (6):
- Germany (6):
  - Department for medical informatics, biometry and epidemiology, Ruhr-University of Bochum, Bochum, North Rhine-Westphalia
  - Institute of Clinical Chemistry, Transfusion and Laboratory Medicine, Universitätsklinikum Bergmannsheil, Ruhr-Universität Bochum, Bochum, North Rhine-Westphalia
  - Medical Hospital II, Bergmannsheil University Hospitals, Ruhr University of Bochum, Bochum, North Rhine-Westphalia
  - Medizinische Klinik I, Universitätsklinikum Bergmannsheil, Ruhr-Universität Bochum, Bochum, North Rhine-Westphalia
  - Diabetes-Zentrum, Mathias-Spital, Rheine, North Rhine-Westphalia
  - Abteilung für Laboratoriums- und Transfusionsmedizin, Westpfalz-Klinikum Kaiserslautern, Kaiserslautern, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dietrich JW, Stachon A, Antic B, Klein HH, Hering S. The AQUA-FONTIS study: protocol of a multidisciplinary, cross-sectional and prospective longitudinal study for developing standardized diagnostics and classification of non-thyroidal illness syndrome. BMC Endocr Disord. 2008 Oct 13;8:13. doi: 10.1186/1472-6823-8-13. PMID 18851740
- [Background] Dietrich JW, Landgrafe G, Fotiadou EH. TSH and Thyrotropic Agonists: Key Actors in Thyroid Homeostasis. J Thyroid Res. 2012;2012:351864. doi: 10.1155/2012/351864. Epub 2012 Dec 30. PMID 23365787
- [Background] Dietrich JW, Muller P, Schiedat F, Schlomicher M, Strauch J, Chatzitomaris A, Klein HH, Mugge A, Kohrle J, Rijntjes E, Lehmphul I. Nonthyroidal Illness Syndrome in Cardiac Illness Involves Elevated Concentrations of 3,5-Diiodothyronine and Correlates with Atrial Remodeling. Eur Thyroid J. 2015 Jun;4(2):129-37. doi: 10.1159/000381543. Epub 2015 May 23. PMID 26279999
- [Background] Dietrich JW, Landgrafe-Mende G, Wiora E, Chatzitomaris A, Klein HH, Midgley JE, Hoermann R. Calculated Parameters of Thyroid Homeostasis: Emerging Tools for Differential Diagnosis and Clinical Research. Front Endocrinol (Lausanne). 2016 Jun 9;7:57. doi: 10.3389/fendo.2016.00057. eCollection 2016. PMID 27375554
- [Background] Chatzitomaris A, Hoermann R, Midgley JE, Hering S, Urban A, Dietrich B, Abood A, Klein HH, Dietrich JW. Thyroid Allostasis-Adaptive Responses of Thyrotropic Feedback Control to Conditions of Strain, Stress, and Developmental Programming. Front Endocrinol (Lausanne). 2017 Jul 20;8:163. doi: 10.3389/fendo.2017.00163. eCollection 2017. PMID 28775711
- [Background] Dietrich JW, Midgley JEM, Hoermann R. Editorial: "Homeostasis and Allostasis of Thyroid Function". Front Endocrinol (Lausanne). 2018 Jun 5;9:287. doi: 10.3389/fendo.2018.00287. eCollection 2018. No abstract available. PMID 29922229
- [Result] Aweimer A, El-Battrawy I, Akin I, Borggrefe M, Mugge A, Patsalis PC, Urban A, Kummer M, Vasileva S, Stachon A, Hering S, Dietrich JW. Abnormal thyroid function is common in takotsubo syndrome and depends on two distinct mechanisms: results of a multicentre observational study. J Intern Med. 2021 May;289(5):675-687. doi: 10.1111/joim.13189. Epub 2020 Nov 12. PMID 33179374
- See also: Public study site — http://www.aqua-fontis.eu